CLINICAL TRIAL: NCT06620666
Title: Improvement of Biological and Functional Longevity Through Advanced Neuromuscular Training Protocols and Resources in Adulthood.
Brief Title: NEUROmuscular Training for Enhanced AGE Longevity
Acronym: NEUROAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Generalitat Valenciana (Other); Indiex Sport Nutrition Spail SL (Unknown)
Responsible Party: Principal Investigator, Juan C. Colado, Distinguished Chaired Full Professor of Physical Education and Sports, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1861154; CIACIF/2021/189 (Other Grant/Funding Number: Department of Education, Culture, Universities, and Employment of the Valencian Government (Spain))
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Aging; Physical Activity; Training
Keywords: Aging; Dose-response; Variable resistance training; Exercise modalities; Exercise intensities; Oxidative stress; Bone health; Neuromuscular physiology; Physical activity; Cellular aging; Training devices; Dietary supplements; Strength training; Cognitive function; Body composition; Metabolic profile; Inflammatory profile; Immunological profile; Physical performance; DNA damage
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: This is a randomized, duoble-blind (sport scientiest assistance/care assistance-outcome assessor), 12 arms prospective parallel design clinical trial. The older adults will be recruited from the researchers setting and will be randomized in a prospective clinical trial study with a 12 parallel arms study design to a resistance training modalities performed at different intensities or a control groups over a 12-16 weeks period.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: For masking the participants, the investigators will not inform participants of what group they will be in. For outcome assessor, data collectors and data analysts independent people will be use, and if this is not possible, a random code will be created for each participant so that it is not possible to identify which group belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Water-based power resistance training + Dietary supplement I (WPowDSI) (Experimental)
  Interventions: Dietary Supplement: Water-based power resistance training + Dietary supplement I (WPowDSI)
- Water-based power resistance training + Placebo (WPowPl) (Active Comparator)
  Interventions: Dietary Supplement: Water-based power resistance training + Placebo (WPowPl)
- Elastic band-based power resistance training + Dietary supplement I (EBPowDSI) (Experimental)
  Interventions: Dietary Supplement: Elastic band-based power resistance training + Dietary supplement I (EBPowDSI)
- Elastic band-based power resistance training + Placebo (EBPowPl) (Active Comparator)
  Interventions: Dietary Supplement: Elastic band-based power resistance training + Placebo (EBPowPl)
- Elastic band-based eccentric resistance training + Dietary supplement II (EBEccDSII) (Experimental)
  Interventions: Dietary Supplement: Elastic band-based eccentric resistance training + Dietary supplement II (EBEccDSII)
- Elastic band-based eccentric resistance training + Placebo (EBEccPl) (Active Comparator)
  Interventions: Dietary Supplement: Elastic band-based eccentric resistance training + Placebo (EBEccPl)
- Elastic band-based maximum strength resistance training + Dietary supplement II (EBMaxDSII) (Experimental)
  Interventions: Dietary Supplement: Elastic band-based maximum strength resistance training + Dietary supplement II (EBMaxDSII)
- Elastic band-based maximum strength resistance training + Placebo (EBMaxPl) (Active Comparator)
  Interventions: Dietary Supplement: Elastic band-based maximum strength resistance training + Placebo (EBMaxPl)
- Control + Dietary supplement I (CDSI) (Active Comparator)
  Interventions: Dietary Supplement: Control + Dietary supplement I (CDSI)
- Control + Dietary supplement II (CDSII) (Active Comparator)
  Interventions: Dietary Supplement: Control + Dietary supplement (CDSII)
- Control + Placebo (CPl) (Placebo Comparator)
  Interventions: Dietary Supplement: Control + Placebo (CPl)
- Aerobic training + Placebo (AerPl) (Active Comparator)
  Interventions: Dietary Supplement: Active Comparator: Aerobic training + Placebo (AerPl)

INTERVENTIONS:
Dietary Supplement: Water-based power resistance training + Dietary supplement I (WPowDSI) — The WPowDSI group will perform 8 repetitions per exercise (arm fly and swing, small and big kick, and a combined upper and lower limb exercise). Regarding the perceived exertion rating, a value of 4 (1º repetition) and 7 (last repetition) was recorded, accorded to an adaptation of the OMNI-RES scale in water in the remaining 12-16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 90s of active recovery (slow rhythmic swinging of the extremities) between sets. The speed of execution of the exercises was controlled using a metronome marking the cadence (concentric phase as fast as possible; eccentric phase 2s). Devices were used according to individual needs. Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Water-based power resistance training + Dietary supplement I (WPowDSI)
Dietary Supplement: Water-based power resistance training + Placebo (WPowPl) — The WPowCr group will perform 8 repetitions per exercise (arm fly and swing, small and big kick, and a combined upper and lower limb exercise). Regarding the perceived exertion rating, a value of 4 (1º repetition) and 7 (last repetition) was recorded, accorded to an adaptation of the OMNI-RES scale in water in the remaining 12-16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 90s of active recovery (slow rhythmic swinging of the extremities) between sets. The speed of execution of the exercises was controlled using a metronome marking the cadence (concentric phase as fast as possible; eccentric phase 2s). Devices were used according to individual needs. Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Water-based power resistance training + Placebo (WPowPl)
Dietary Supplement: Elastic band-based power resistance training + Dietary supplement I (EBPowDSI) — The EBPowDSI group will perform 8 repetitions per exercise (militar press, squat, upright row, lunge, and push-press). Regarding the perceived exertion rating, a value of 4 (1º repetition) and 7 (last repetition), according to an adaptation of the OMNI-RES EB scale in the remaining 12-16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 90s of active recovery (slow rhythmic swinging of the extremities) between sets and 90s of rest between exercises. The speed of execution of the exercises was controlled using a metronome marking the cadence (concentric phase: as fast as possible; eccentric phase: 2s). Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based power resistance training + Dietary supplement I (EBPowDSI)
Dietary Supplement: Elastic band-based power resistance training + Placebo (EBPowPl) — The EBPotPl group will perform 8 repetitions per exercise (militar press, squat, upright row, lunge, and push-press). Regarding the perceived exertion rating, a value of 4 (1º repetition,) and 7 (last repetition), according to an adaptation of the OMNI-RES EB scale in the remaining 16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 90s of active recovery (slow rhythmic swinging of the extremities) between sets and 90s of rest between exercises. The speed of execution of the exercises was controlled using a metronome marking the cadence (concentric phase: as fast as possible; eccentric phase: 2s). Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based power resistance training + Placebo (EBPowPl)
Dietary Supplement: Elastic band-based eccentric resistance training + Dietary supplement II (EBEccDSII) — The EBEccDSII group will perform 6 repetitions per exercise (lunge, chest press, hiptrust and standing row). The exercises were performed at maximum intensity until the point where stability or technique was lost, prior the stretching of the band. The number of sets throughout the entire intervention was 4 sets per exercise, with 120s of active recovery between sets and 90s of rest between exercises. The pace of execution of the exercises was controlled using a metronome marking the cadence (concentric phase: until reaching the stretching of the band; eccentric phase: 5s). Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based eccentric resistance training + Dietary supplement II (EBEccDSII)
Dietary Supplement: Elastic band-based eccentric resistance training + Placebo (EBEccPl) — The EBEccPl group will perform 6 repetitions per exercise (lunge, chest press, hiptrust and standing row). The exercises were performed at maximum intensity until the point where stability or technique was lost, prior the stretching of the band. The number of sets throughout the entire intervention was 4 sets per exercise, with 120s of active recovery between sets and 90s of rest between exercises. The pace of execution of the exercises was controlled using a metronome marking the cadence (concentric phase: until reaching the stretching of the band; eccentric phase: 5s). Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based eccentric resistance training + Placebo (EBEccPl)
Dietary Supplement: Elastic band-based maximum strength resistance training + Dietary supplement II (EBMaxDSII) — The EBMaxDSII group will perform 6 repetitions per exercise (lunge, chest press, hiptrust and standing row). Regarding the perceived exertion rating, a value of 7 (1º repetition,) and 9 (last repetition), according to an adaptation of the OMNI-RES EB scale in the remaining 16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 120s of active recovery between sets and 90s of rest between exercises. The pace of execution of the exercises was controlled using a metronome marking the cadence (concentric-eccentric phase: 2s). Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based maximum strength resistance training + Dietary supplement II (EBMaxDSII)
Dietary Supplement: Elastic band-based maximum strength resistance training + Placebo (EBMaxPl) — The EBMaxPl group will perform 6 repetitions per exercise (lunge, chest press, hiptrust and standing row). Regarding the perceived exertion rating, a value of 7 (1º repetition,) and 9 (last repetition), according to an adaptation of the OMNI-RES EB scale in the remaining 16 weeks. The number of sets throughout the entire intervention was 4 sets per exercise, with 120s of active recovery between sets and 90s of rest between exercises. The pace of execution of the exercises was controlled using a metronome marking the cadence (concentric-eccentric phase: 2s). Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Elastic band-based maximum strength resistance training + Placebo (EBMaxPl)
Dietary Supplement: Control + Placebo (CPl) — Participants randomized into the control group will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet. Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Control + Placebo (CPl)
Dietary Supplement: Control + Dietary supplement I (CDSI) — Participants randomized into the control group will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet. Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Control + Dietary supplement I (CDSI)
Dietary Supplement: Control + Dietary supplement (CDSII) — Participants randomized into the control group will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet. Regarding supplementation, participants were randomly assigned to receive their daily dose.
  Arms: Control + Dietary supplement II (CDSII)
Dietary Supplement: Active Comparator: Aerobic training + Placebo (AerPl) — The group will perform aerobic exercise for 20-40 minutes with easy execution exercise. Regarding placebo, participants were randomly assigned to receive their daily dose.
  Arms: Aerobic training + Placebo (AerPl)

SUMMARY:
In recent years the research group on Prevention and Health in Exercise and Sport (PHES) has carried out numerous studies that have provided current and convincing evidence of the benefits of physical activity and exercise for chronic health, but unfortunately it has also shown that if physical exercise is not properly prescribed it can impair health, as well as accelerating the ageing process.

The research proposal presented here aims to reveal some of the forms of physical exercise and resources for its application that may be most beneficial for people's health, thus trying to find reliable evidence that will increase healthy longevity and quality of life in society.

Based on the above, and taking into account that the possible beneficial adaptations for health are specific to the applied form of physical exercise and the equipment used during its development, the PHES research group wishes to investigate the most appropriate strategies to ensure an active and positive ageing process.

With these relevant findings the researchers can create specific action plans for prevention and promotion through physical exercise in order to improve both health and quality of life expectancy.

The general objective of the project is to identify the most advanced methods and material resources with which to guarantee a beneficial process of active and healthy ageing with chronic training, so that with these relevant findings, concrete action plans can be created for prevention and promotion through physical exercise in order to improve both health and quality of life expectancy.

The specific objectives are the following:

* To validate new, specific, safe, and efficient tools to monitor the intensity of neuromuscular strength training activities in older adults.
* To analyze and compare the chronic effects of different cardiovascular and neuromuscular strength training modalities applied with different materials on cellular ageing, body composition, metabolic, and immune profiles, cognitive function, motor function, quality of life and well-being in older adults.
* To evaluate the efficacy of the use of dietary supplements to reduce or even stop the chronic adverse effects that different physical activity levels and/or physical exercise programs can have on the oxidative and inflammatory profile, body composition and metabolic profile, muscle and DNA damage, and physical performance in older adults.

DETAILED DESCRIPTION:
The project presented here will consist of two stages:

(i) Stage 1 "Validation studies": They consist in the development of validation of perceptual tools for pre-exercise quantification of the intensity of the training protocols with different training materials and methodologies; The research in this first stage will take the form of a descriptive cross-sectional perceptual estimation studies. Therefore, this first stage of research will be performed prior to the application of the chronic studies, and they will focus on validating resources for the proper control of intensity during the application of resistance training in elderly individuals by using measures of pre-exercise perceived exertion. If these concepts are validated, the researchers could state that will have created easily applicable and universal tools that will help to extend the appropriate use resistance training in older adults with highly accessible materials and conditions that can be applied internationally.

(ii) Stage 2 "Chronic studies": They consist in the development of different intervention protocols to analyze the chronic effects of different regime of methodologies, materials, and food supplementation. The research project presented here will continue in these second stages with prospective experimental studies of randomized intervention with older adults with pre-, and post-treatment measurements. The study population will be older adults belonging to a convenience sample who will participate voluntarily. The study at this stage will consist of carrying out different intervention protocols over a period of 12-16 weeks.

All the training programs of the chronic studies will start with familiarization sessions. During the first familiarization sessions, participants will be instructed on how to obtain the measure of the perceived exertion scale appropriate to the exercise intensity to be developed and also how to correctly perform the exercises of the training program. As for the training plan, in the different experimental groups, participants will complete a list of exercises prescribed by the technicians, which will be repeated in each session throughout the training plan. Participants assigned to the sedentary control groups will be asked to continue with their normal diet and activities during the weeks of the study and will be prohibited from participating in any physical activity program or weight loss plan. In contrast, the experimental groups will perform a strength training program with the modality-specific method developed and with the type of material and/or dietary supplement that corresponds to them according to the experimental design at a frequency of 2-3 days per week for 12-16 weeks. The standard exercise session will have a protocolized structure with a warm-up, a main exercise part and a cool-down.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults (≥ 60 years), i.e., no physical exercise.
* Physically independent (able to walk 100 m without a walking aid and climb 10 steps without rest).
* Medical certificate of suitability or fitness to practice resistance training activities.
* Cognitive ability to understand and follow the instructions and sign the informed consent form.
* Free of any antioxidant supplements for at least six weeks before the start of this study: Vitamin C, Vitamin E, Vitamin A (beta-carotene), Zinc, Coenzyme Q (CoenzymeQ10), turmeric, Omega 3, creatine monohydrate or multivitamin products containing any of these compounds.
* Do not smoke more than 5 cigarettes per day or consume distilled alcoholic beverages on a daily basis.

Exclusion Criteria:

* Presence of cardiovascular, musculoskeletal, renal, liver, pulmonary, or neuromuscular and neurological disorders that would prevent the participant from performing the exercises.
* A history of malignant neoplasms.
* Terminal illness with life expectancy of less than one year.
* Mini mental State Examination lower than 23/30.
* Severe visual or hearing impairment.
* Body weight changes at 10% in the previous year.
* Intake of prescription medications or supplements (e.g., vitamins C, E) that were expected to alter the results of the study (ergogenic, dietary aids, estrogen, beta-blockers, steroid hormones, calcitonin, corticosteroids, glucocorticoids, thiazide diuretics, anticonvulsants, bisphosphonates, raloxifene).
* Current or prior (past six months) use of hormone replacement therapy.
* Engagement in regular strength training (more than once a week) during the previous six months.
* Participation in another research project (within the last six months) involving dietary, exercise, and/or pharmaceutical intervention.
* Not be under pharmacological treatment with allopurinol (trade name Zyloric).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in lipid peroxidation | Baseline and 12-16 weeks
  The lipid peroxidation will be assessed via blood collections of 8-isoprostaglandin (nmol /mmol)
Change in antioxidants enzymes | Baseline and 12-16 weeks
  The antioxidants enzymes will be assessed via blood collections of glutathione peroxidase (IU/g Hb).
Change in brain neuroplasticity | Baseline and 12-16 weeks
  The brain neuroplasticity will be assessed via blood collections of brain-derived neurotrophic factor (BDNF) (ng/ml)
Change in inflammatory profile | Baseline and 12-16 weeks
  The interleukin 6 (IL-6), and tumor necrosis factor alpha (TNF-α) (pg/mL) will be assessed via blood collections.
Change in bone metabolism I (Formation) | Baseline and 12-16 weeks
  The bone metabolism will be assessed via blood collections of Type I procollagen N-terminal propeptide (P1NP) are marker of bone formation.
Change in bone metabolism II (Resorption) | Baseline and 12-16 weeks
  The bone metabolism will be assessed via blood collections of terminal telopeptide of collagen type I (β-CTX- 1) which is a marker of bone resoption.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and 12-16 weeks
  Systolic and diastolic blood pressure (mmHg) will be measured
Change in renal and hepatic profile I | Baseline and 12-16 weeks
  Glutamic-oxaloacetic transaminase (U/L) will be measured.
Change in renal and hepatic profile II | Baseline and 12-16 weeks
  Creatine (mg/dL) will be measured.
Change in lipid profile | Baseline and 12-16 weeks
  The lipid profile will be assessed via blood collections: total cholesterol (mg/dL), high-density lipoprotein cholesterol (mg/dL), low-density lipoprotein cholesterol (mg/dL) and triglycerides (mg/dL).
Change in metabolic profile I | Baseline and 12-16 weeks
  The metabolic profile will be assessed via blood collections of basal glucose (mmol/l).
Change in metabolic profile II | Baseline and 12-16 weeks
  The metabolic profile will be assessed via blood collections of human ghrelin (GHRL) (pg/ml), human acylated ghrelin (AG) (pg/ml), human glucagon like peptide 1 (GLP1) (pg/ml), and human cholecystokinin (CCK) (pg/ml).
Change in metabolic profile III | Baseline and 12-16 weeks
  The metabolic profile will be assessed via blood collections of leptin (ng/mL).
Change in metabolic profile IV | Baseline and 12-16 weeks
  The metabolic profile will be assessed via blood collections of human peptide YY (PYY) (10 µCi).
Change in cognitive function I | Baseline and 12-16 weeks
  The cognitive function will be assessed by the Trail Making Test (TMT) questionnaire (seconds; mistakes).
Change in cognitive function II | Baseline and 12-16 weeks
  It will be assessed through the application of the MMSE. This test evaluates cognitive impairment, it contains 28 closed questions that measure 8 of the 11 main aspects of cognitive status.
Change in cognitive function III | Baseline and 12-16 weeks
  It will be measured by Wisconsin Card Sorting Test (WCST). This test measures abstraction ability, concept formation, and cognitive strategy change in response to changes in environmental contingencies.
Change in cognitive function IV | Baseline and 12-16 weeks
  It will be measured by Vienna Test System (VTS). Specifically, will be use the Determination Test (DT), and Reaction Test (RT). This tests are used to check the capacity of observation and visual control, as well as the visual capacity of orientation and the speed of comprehension.

OTHER OUTCOMES:
Change in isokinetic muscle strength | Baseline and 12-16 weeks
  The dynamic maximal concentric muscle strength of the dominant side of knee, elbow, and shoulder (flexion and extension muscle groups) will be measured with an isokinetic dynamometer (Biodex System 4 Pro; Biodex, Shirley, NY) at two angular velocities, 60°/s and 180°/s. Maximal voluntary concentric isokinetic torque will be assessed in Newton-meters (N-m).
Change in maximal muscle hand grip strength | Baseline and 12-16 weeks
  The isometric maximal muscle hand grip strength of both hands will be measured with a dynamometer (kg).
Change in fracture risk | Baseline and 12-16 weeks
  Will be assessed via the FRAX ® tool (%).
Change T-Score | Baseline and 12-16 weeks
  T-Score (SD) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Wards triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in bone mineral density (BMD) | Baseline and 12-16 weeks
  BMD (g/cm2) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Wards triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change bone mineral content (BMC) | Baseline and 12-16 weeks
  BMC(g) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Wards triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in self-reported quality of life | Baseline and 12-16 weeks
  Will be assessed via Short form quality of life questionnaire (SF36) (0-100 points).
State of instrumental activities of daily living | Baseline
  Will be assessed via Lawton and Brody instrumental activities of daily living scale. There are eight domains of function measured with the Lawton and Brody scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
State of basic activities of daily living | Baseline
  Will be assessed via Barthel index of activities of daily living (score 0-100).
Attendance to training program | 12-16 weeks
  Adherence levels (%) will be calculated at the end of the training period. Nonadherence is define as those not attending at follow-up and have not attend for 4 weeks during the training period, and have not given a reason for nonattendance or those who have stated they are dropping out.
State of eye health I | Baseline and 12-16 weeks
  The eye health will be measured with Visual Function index (VF14) (0-100 points). This test provides an subjective assessment of visual quality.
State of eye health II | Baseline and 12-16 weeks
  The state of eye health will be measured with Functional Acuity Contrast Test (FACT) (log) associated with contrast sensitivity.
State of eye health III | Baseline and 12-16 weeks
  The intraocular pressure will be measured using an iCare rebound tonometer (mmHg).
State of eye health IV | Baseline and 12-16 weeks
  The ocular perfusion pressure (mmHg) will be calculate with a formula that includes intraocular pressure and blood pressure.
Change in neuropathic pain I | Baseline and 12-16 weeks
  Neuropathic pain will be measured with Western Ontario and McMaster Universities Arthritis Index (WOMAC). This index is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: a) pain (0-20 points); b) stiffness (0-8 points); c) physical function (0-68 points).
Change in neuropathic pain II | Baseline and 12-16 weeks
  Neuropathic pain will be measured with Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale. This scale can be used to identify pain of predominantly neuropathic origin, thus distinguishing between neuropathic pain and nociceptive pain. The LANSS scale comprises of a 7-item pain scale (5 are symptom related, and 2 are examination items) (more than 12 points on the scale might also be suffering from neuropathic pain; less than 12 points on the scale might not be suffering from neuropathic pain).
Change in neuropathic pain III | Baseline and 12-16 weeks
  Neuropathic pain will be measured with Visual Analogue Scale (VAS) scale. This scale measure the intensity or frequency of various symptoms (0-100 points; A higher score indicates greater pain intensity).
Change in neuropathic pain IV | Baseline and 12-16 weeks
  Neuropathic pain will be measured with Neuropathic pain scale (NPS). This scale measures 10 specific qualities associated with neuropathic pain (0-10 points; A higher score indicates greater pain intensity).
Height | Baseline and 12-16 weeks
  Height (cm) will be recorded to the nearest 0.01 cm using a stadiometer (Seca 711, Hamburg, Germany)
Weight | Baseline and 12-16 weeks
  Weight (kg) will be measured with a bioelectrical impedance scale (Tanita model Tanita MC 780-P MA, Tokyo, Japan; precision 0.01 kg).
Body Mass Index | Baseline and 12-16 weeks
  Weight and height will be combined to report body mass index (BMI) (kg/m^2 ).
Change in body composition I (Fat mass) | Baseline and 12-16 weeks
  Fat mass (kg) will be assessed for whole body and appendicular/visceral regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA). Furthermore, the same variable will be assessed using a bioelectrical impedance scale (Tanita model Tanita MC 780-P MA, Tokyo, Japan; precision 0.01 kg).
Change in body composition II (% Fat mass) | Baseline and 12-16 weeks
  Percentage of fat mass (%) will be assessed for whole body and appendicular/visceral regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA). Furthermore, the same variable will be assessed using a bioelectrical impedance scale (Tanita model Tanita MC 780-P MA, Tokyo, Japan; precision 0.01 kg).
Change in body composition III (Fat-free mass) | Baseline and 12-16 weeks
  Fat-free mass (kg) will be assessed for whole body and appendicular/visceral regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA). Furthermore, the same variable will be assessed using a bioelectrical impedance scale (Tanita model MC 780-P MA, Tokyo, Japan; precision 0.01 kg).
State of nutritional status | Baseline and 12-16 weeks
  Dietary intake will be assessed by applying the Mini Nutritional Assessment-short form (MNA-f1). This brief questionnaire consists of six items, which correspond to questions about decreased food consumption, weight loss, mobility, presence of acute illness, neuropsychological problems and anthropometry.
Change in balance I | Baseline and 12-16 weeks
  Balance will be measured with Romberg test (points).
Change in balance II | Baseline and 12-16 weeks
  Balance will be measured with Functional Reach Test (FRT) (cm).
Change in functional performance I | Baseline and 12-16 weeks
  The functional performance will be assessed with Senior Fitness tests that involve 3 tests: Chair Stand (stand up from a chair as often as possible within 30s); Up-and-Go (for dynamic balance, time for got up from the chair, walk as quickly as possible around a cone placed 2.4 m from the chair, and resume the seated position); and Six-Minute walking test (for aerobic capacity, distance walked in 6 minutes).
Change in functional performance II | Baseline and 12-16 weeks
  It will be measured by Short Physical Performance Battery (SPPB): This is a performance instrument that includes 3 tests: balance, walking speed and getting up and sitting down from a chair 5 times. Each test is scored from 0 (worst performance) to 4 (best performance). A total score is obtained for the entire battery, which is the sum of the 3 tests and ranges from 0 to 12 and is classified as: low performance (0-6 points); intermediate (7-9 points) and high performance (10-12 points)
Change in functional performance III | Baseline and 12-16 weeks
  It will be measured by 2-Minute Step Test: The test considers the number of times the right knee reaches the individual reference height. If it does not reach the indicated height, the speed will be reduced so that the test is valid without stopping time. The score at the end will be given according to the number of steps taken, where the right knee reached the set height.
Change in depressive symptoms | Baseline and 12-16 weeks
  It will be measured through the GDS-15 test, the most widely used screening scale for depression in older people, consisting of 15 questions, with a dichotomous yes/no response. Scores from 0 to 4 points are considered normal, 5-10 indicates mild depression, and scores greater than 10 indicate established depression
State of level of physical activity I | Baseline and 12-16 weeks
  The level of physical activity (low, medium, high) of the participants will be assessed by Global Physical Activity Questionnaire (GPAQ) (min/week; MET/week).
State of level of physical activity II | Baseline and 12-16 weeks
  The level of physical activity (low, medium, high) of the participants will be assessed by International Physical Activity Questionnaires (IPAQ) (min/week; MET/week).
Working heart rate | Baseline and 12-16 weeks
  Working heart rate will be assessed with a Polar FT1 (Polar Electro, Tampere, Finland) (bpm). This variable will be measured in the first stage of the project (Validation studies.
Neuromuscular activation | Baseline and 4 weeks
  Neuromuscular activation will be measured using electromyographic (EMG). The EMG signal will be obtained using two two-channel handheld devices (RealtimeTechnologies Ltd., Dublin, Ireland) with 16-bit analog-to-digital (A/D) conversion. EMGdata will be monitored using validated mDurance software for Android (mDuranceSolutions S.L., Granada, Spain). This variable will be measured in the first stage of the project (Validation studies).
Total repetitions performed | Baseline and 4 weeks
  Total repetitions performed will be recorded for later analysis with photogrammetry and video techniques. This variable will be measured in the first stage of the project (Validation studies).
Maximum oxygen consumption | Baseline and 4 weeks
  Will be measured using a portable metabolimeter (VO2 Master Health Sensors Inc., Canada) (ml/kg/min).
Capillary blood lactate | Baseline and 4 weeks
  Blood lactate concentrations will be measured from capillary blood obtained from the fingertips. The samples were analyzed using a portablel actate analyzer (Lactate Pro 2, Arkray Inc., Kyoto, Japan) (mmol/L).
Rating of perceived exertion | Baseline and 4 weeks
  Rating of perceived exertion will be measured with OMNI-Resistance Exercise Scale in the elderly (0-10 points). This variable will be measured in the first stage of the project (Validation studies).
Change in sleep quality | Baseline and 12-16 weeks
  It will be assessed by the Pittsburgh Sleep Quality Questionnaire. This instrument provides an overall score of subjects sleep quality and 7 partial scores belonging to different partial scores pertaining to different components: subjective sleep quality, latency, duration, habitual efficiency, disturbances, use of hypnotic medication and daytime dysfunction. The questions refer to the last month. The score for each of the seven components ranges from 0 (no difficulty) to 3 (severe difficulty); the overall score ranges between 0 (no difficulty) and 21 (difficulties in all areas), with a cut-off point at score 5 to differentiate between good and bad sleepers.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Activity and Sport Science Faculty, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No